CLINICAL TRIAL: NCT00732225
Title: A Prospective, Non-randomized Comparison of DisCoVisc to Dispersive and Cohesive Ophthalmic Viscosurgical Devices (OVDs) in Non-eventful Cataract Surgery
Brief Title: DisCoVisc Comparative Evaluation
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Alcon Research (Industry)
Responsible Party: Rick Potvin/Director - Global Scientific Market Affairs, Alcon Research
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: M07-015
Record Dates: First submitted 2008-08-07; First posted 2008-08-11 (Estimated); Results first posted 2010-07-30 (Estimated); Last update posted 2010-07-30 (Estimated); Status verified 2010-06

CONDITIONS: Cataracts
Keywords: DisCoVisc OVD; Ophthalmic Viscosurgical Device
MeSH Terms: conditions — Cataract

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (5):
- DisCoVisc (Active Comparator): Alcon DisCoVisc Ophthalmic Viscosurgical Device (OVD) (4% sodium chondroitin sulfate, 1.65% sodium hyaluronate)
  Interventions: Device: DisCoVisc
- DuoVisc (Active Comparator): Alcon DuoVisc Ophthalmic Viscosurgical System (1% sodium hyaluronate, and 3% sodium hyaluronate, 4% chondroitin sulfate)
  Interventions: Device: DuoVisc
- BioVisc (Active Comparator): Sophia Lab BioVisc Ophthalmic Viscosurgical Device (OVD) (1% sodium hyaluronate)
  Interventions: Device: BioVisc
- Healon5 (Active Comparator): AMO Healon5 Ophthalmic Viscosurgical Device (OVD) (2.3% Sodium Hyaluronate)
  Interventions: Device: Healon5
- Amvisc Plus (Active Comparator): Bausch & Lomb Amvisc Plus Ophthalmic Viscosurgical Device (OVD) (1.6% Sodium Hyaluronate)
  Interventions: Device: Amvisc Plus

INTERVENTIONS:
Device: DisCoVisc — DisCoVisc Ophthalmic Viscosurgical Device (OVD) (4% sodium chondroitin sulfate, 1.65% sodium hyaluronate) as utilized throughout cataract removal and intraocular lens (IOL) insertion procedure.
  Arms: DisCoVisc
Device: DuoVisc — DuoVisc Ophthalmic Viscosurgical System (1% sodium hyaluronate, and 3% sodium hyaluronate, 4% chondroitin sulfate) as utilized throughout cataract removal and intraocular lens (IOL) insertion procedure.
  Arms: DuoVisc
Device: BioVisc — BioVisc Ophthalmic Viscosurgical Device (OVD) (1% sodium hyaluronate) as utilized throughout cataract removal and intraocular lens (IOL) insertion procedure.
  Arms: BioVisc
Device: Healon5 — Healon5 Ophthalmic Viscosurgical Device (OVD) (2.3% Sodium Hyaluronate) as utilized throughout cataract removal and intraocular lens (IOL) insertion procedure.
  Arms: Healon5
Device: Amvisc Plus — Amvisc Plus Ophthalmic Viscosurgical Device (OVD) (1.6% Sodium Hyaluronate) as utilized throughout cataract removal and intraocular lens (IOL) insertion procedure.
  Arms: Amvisc Plus

SUMMARY:
A comparison of the ability of DisCoVisc to that of other Opthalmic Viscosurgical Devices (OVDs) (DuoVisc®, BioVisc®, Healon5®, or Amvisc PLUS) regarding endothelial protection and anterior chamber space maintenance during non-eventful cataract surgery.

ELIGIBILITY:
Inclusion Criteria:

* Unilateral operable cataracts

Exclusion Criteria:

* Preoperative Endothelial Cell Count (ECC) ≤1500 cells/mm2
* Intraocular Pressure (IOP) > 21
* History of ocular inflammation
* Systemic or ocular diseases affecting corneal endothelium

Min Age: 49 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 173 (Actual)
Dates: Start 2007-05; Primary Completion 2008-02 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Alcon Call Center for Trial Locations, Fort Worth, Texas, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Preoperatively, subjects were examined to ensure they met the inclusion/exclusion criteria. Patients were >49 years of age, of any race and either gender. Patients had operable cataracts in at least one eye and were able to provide informed consent
Pre-assignment Details: As access to Ophthalmic Viscosurgical Devices (OVDs) was limited, patients received whichever OVD was in stock at the time of surgery. 51 patients had a different OVD used in each eye. As a result, their demographic data is included in 2 OVD groups, resulting in a total of 224 patients (when group totals are added).
Groups:
- AmviscPlus: Bausch & Lomb AmviscPlus Ophthalmic Viscosurgical Device (OVD) (1.6% Sodium Hyaluronate)
Period: Overall Study
Arm/Group | DisCoVisc | DuoVisc | BioVisc | Healon5 | AmviscPlus
Started | 71 (76 eyes of 71 patients) | 40 (41 eyes of 40 patients) | 26 (26 eyes of 26 patients) | 33 (33 eyes of 33 patients) | 54 (55 eyes of 54 patients)
Completed | 60 (64 eyes of 60 patients) | 32 (33 eyes of 32 patients) | 23 (23 eyes of 23 patients) | 29 (29 eyes of 29 patients) | 48 (48 eyes of 48 patients)
Not Completed | 11 | 8 | 3 | 4 | 6

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | DisCoVisc | DuoVisc | BioVisc | Healon5 | AmviscPlus | Total
Number analyzed (Participants) | 71 | 40 | 26 | 33 | 54 | 224
Age Continuous [Mean (Standard Deviation); unit: years] — Age not available for the following: 7 Discovisc patients, 11 Duovisc patients, 3 Biovisc patients, 4 Amvisc Plus patients. Total mean age and standard deviation not calculated.
  years | 66.8 (9.54) | 67.31 (12.61) | 71.48 (8.56) | 67.03 (12.13) | 66.24 (10.51) | 67.9 (10.8)
Gender [Number; unit: participants] — Gender not available for the following: 2 Discovisc patients, 2 Duovisc patients, 1 Biovisc patient, 2 Amvisc Plus patients.
  participants
    Female | 42 | 22 | 13 | 19 | 29 | 125
    Male | 27 | 16 | 12 | 14 | 23 | 92

OUTCOME MEASURES:

1. Primary Outcome: Percent Loss of Endothelial Cells
Description: Percentage of corneal endothelial cells lost 2 months after surgery as compared to the number of corneal endothelial cells measured before the operation. Corneal Endothelial Cells are measured by counting the number of cells on an image taken by specular microscope.
Time Frame: 2 months following surgery
Population: This data was collected on the eyes of patients attending the visit 2 months after surgery.
Measure: Mean (Standard Deviation); unit: Percent Loss
Arm/Group | DisCoVisc | DuoVisc | BioVisc | Healon5 | AmviscPlus
Number analyzed (Participants) | 64 | 32 | 23 | 29 | 46
Percent Loss | 9.48 (20.72) | 15.66 (11.03) | 23.69 (13.47) | 25.70 (13.94) | 23.04 (16.20)

2. Secondary Outcome: Aqueous Signs - Corneal Edema
Description: Measured as the percentage of patient's eyes subjectively evaluated to have corneal edema at each of the following gradings:
  0 - None
  1. - Mild, slight localized or generalized edema
  2. - Moderate, significant localized or generalized edema
  3. - Severe, advanced localized or generalized edema
Time Frame: 1 day after surgery
Population: This data was collected on all eyes of patients attending the 1-day visit.
Measure: Number; unit: Percentage of Eyes
Arm/Group | DisCoVisc | DuoVisc | BioVisc | Healon5 | AmviscPlus
Number analyzed (Participants) | 75 | 41 | 24 | 33 | 55
Percentage of Eyes
  None | 81.33 | 78.05 | 37.50 | 63.64 | 54.55
  Mild | 14.67 | 19.51 | 37.50 | 30.30 | 32.73
  Moderate | 4.00 | 2.44 | 25.00 | 6.06 | 12.73
  Severe | 0.00 | 0.00 | 0.00 | 0.00 | 0.00

3. Secondary Outcome: Aqueous Signs - Aqueous Flare
Description: Measured as the percentage of patient's eyes subjectively evaluated to have Aqueous Flare at each of the following gradings:
  0-None: No visible flare when compared with the normal eye.
  1. Mild: Flare visible against dark papillary background but not visible against iris background.
  2. Moderate: Flare is visible with the slit-lamp beam aimed onto the iris surface as well as the dark papillary background.
  3. Severe: Very dense flare. May also present as a hazy appearance of anterior segment structures when viewed with low power magnification of the slit-lamp.
Time Frame: 1 day following surgery
Population: This data was collected on all eyes of patients attending the 1 day postoperative visit.
Measure: Number; unit: Percentage of Eyes
Arm/Group | DisCoVisc | DuoVisc | BioVisc | Healon5 | AmviscPlus
Number analyzed (Participants) | 75 | 41 | 24 | 33 | 55
Percentage of Eyes
  None | 76.00 | 75.61 | 41.67 | 63.64 | 54.55
  Mild | 21.33 | 19.51 | 33.33 | 24.24 | 34.55
  Moderate | 2.67 | 4.88 | 25.00 | 12.12 | 10.91
  Severe | 0.00 | 0.00 | 0.00 | 0.00 | 0.00

4. Secondary Outcome: Aqueous Signs - Aqueous Cells
Description: Measured as the percentage of patient's eyes subjectively evaluated to have Aqueous Cells at each of the following gradings:
  0 - None
  1. - 1 to 5 cells
  2. - 6 to 15 cells
  3. - 16 to 30 cells
  4. - >30 cells
Time Frame: 1 day following surgery
Population: This data was collected on all eyes of patients attending the 1 day post-operative visit.
Measure: Number; unit: Percentage of Eyes
Arm/Group | DisCoVisc | DuoVisc | BioVisc | Healon5 | AmviscPlus
Number analyzed (Participants) | 75 | 41 | 24 | 33 | 55
Percentage of Eyes
  Grade 0 | 84.00 | 80.49 | 45.83 | 63.64 | 56.36
  Grade 1 | 16.00 | 17.07 | 25.00 | 27.27 | 36.36
  Grade 2 | 0.00 | 2.44 | 29.17 | 9.09 | 7.27
  Grade 3 | 0.00 | 0.00 | 0.00 | 0.00 | 0.00
  Grade 4 | 0.00 | 0.00 | 0.00 | 0.00 | 0.00

5. Secondary Outcome: Intraocular Pressure (IOP)
Description: Measure of intraocular pressure of a patient's eye via tonometry one day after surgery. Measured in mmHg. Normal intraocular pressure between 10 mmHg and 20 mmHg.
Time Frame: 1 day following surgery
Population: This data was collected on all eyes of patients attending the 1 day postoperative visit with the exception of the following: 3 DisCoVisc patients, 4 DuoVisc patients, 1 Healon5 patient, and 4 Amvisc Plus patients.
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | DisCoVisc | DuoVisc | BioVisc | Healon5 | AmviscPlus
Number analyzed (Participants) | 72 | 37 | 25 | 32 | 51
mmHg | 17.67 (3.88) | 17.78 (3.81) | 20.32 (7.39) | 19.88 (8.90) | 16.96 (4.76)

6. Secondary Outcome: Physician Survey - Anterior Chamber Dome Maintenance During Anterior Capsulotomy
Description: Surgeon reporting of Anterior Chamber Dome Maintenance of a patient's eye During Anterior Capsulotomy. Evaluated on a subjective scale and reported as percent by response. The following scale is used, from worst to best: Flat, Shallow, Working Space Adequate, Full Chamber Maintenance.
Time Frame: Time of Surgery
Population: This data was collected on all eyes of patients undergoing surgery with the exception of the following: 2 DisCoVisc eyes and 2 Healon5 eyes
Measure: Number; unit: Percentage of Eyes
Arm/Group | DisCoVisc | DuoVisc | BioVisc | Healon5 | AmviscPlus
Number analyzed (Participants) | 74 | 41 | 25 | 33 | 55
Percentage of Eyes
  Flat | 0.00 | 0.00 | 0.00 | 0.00 | 0.00
  Shallow | 2.70 | 0.00 | 100.00 | 9.09 | 85.45
  Working Space Adequate | 13.51 | 0.00 | 0.00 | 0.00 | 3.64
  Full Chamber Maintenance | 83.78 | 100.00 | 0.00 | 90.91 | 10.91

7. Secondary Outcome: Physician Survey - Anterior Chamber Dome Maintenance During Phacoemulsification
Description: Surgeon reporting of Anterior Chamber Dome Maintenance of a patient's eye during Phacoemulsification. Evaluated on a subjective scale and reported as percent by response. The following scale is used, from worst to best: Flat, Shallow, Working Space Adequate, Full Chamber Maintenance
Time Frame: Time of Surgery
Population: This data was collected on all eyes of patients undergoing surgery with the exception of the following: 17 DisCoVisc eyes, 19 DuoVisc eyes, 6 BioVisc eyes,3 Healon5 eyes, and 11 Amvisc Plus eyes.
Measure: Number; unit: Percentage of Eyes
Arm/Group | DisCoVisc | DuoVisc | BioVisc | Healon5 | AmviscPlus
Number analyzed (Participants) | 59 | 22 | 20 | 30 | 42
Percentage of Eyes
  Flat | 0.00 | 0.0 | 0.00 | 0.00 | 0.00
  Shallow | 0.00 | 0.00 | 25.00 | 0.00 | 2.38
  Working Space Adequate | 10.17 | 9.09 | 70.00 | 36.67 | 80.95
  Full Chamber Maintenance | 89.83 | 90.91 | 5.00 | 63.33 | 16.67

8. Secondary Outcome: Physician Survey - Anterior Chamber Dome Maintenance During IOL Insertion
Description: Surgeon reporting of Anterior Chamber Dome Maintenance During Intraocular Lens (IOL) insertion into a patient's eye. Evaluated on a subjective scale and reported as percent by response. The scale, from worst to best, is as follows: Flat, Shallow, Working Space Adequate, Full Chamber Maintenance
Time Frame: Time of Surgery
Population: This data was collected on all eyes of patients undergoing surgery with the exception of the following: 17 DisCoVisc eyes, 20 DuoVisc eyes, 6 BioVisc eyes,4 Healon5 eyes, and 14 Amvisc Plus eyes.
Measure: Number; unit: Percentage of Eyes
Arm/Group | DisCoVisc | DuoVisc | BioVisc | Healon5 | AmviscPlus
Number analyzed (Participants) | 59 | 21 | 20 | 29 | 41
Percentage of Eyes
  Flat | 0.00 | 0.00 | 0.00 | 0.00 | 0.00
  Shallow | 0.00 | 0.00 | 10.00 | 0.00 | 4.88
  Working Chamber Adequate | 3.39 | 9.52 | 90.00 | 24.14 | 68.29
  Full Chamber Maintenance | 96.61 | 90.48 | 0.00 | 75.86 | 26.83

ADVERSE EVENTS:
Description: Adverse events collected against the total number of eyes that could be affected instead of patients.
Arm/Group | DisCoVisc | DuoVisc | BioVisc | Healon5 | AmviscPlus
Serious Adverse Events (participants affected / at risk) | 0/76 | 0/41 | 0/26 | 0/33 | 0/55
Other Adverse Events (participants affected / at risk) | 0/76 | 0/41 | 0/26 | 0/33 | 0/55

LIMITATIONS AND CAVEATS:
At the time of surgery, patients were assigned to a study group based on the availability of study Ophthalmic Viscosurgical Devices (OVDs).

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
No paper that incorporates Sponsor Confidential Information will be submitted for publication without Sponsor's prior written agreement.